CLINICAL TRIAL: NCT01158911
Title: Does Uric Acid Promote Progression of Kidney Disease and Development of Cardiovascular Disease in Patients With Chronic Kidney Disease?
Brief Title: Uric Acid and Long-term Outcomes in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Mark Sarnak, MD, Tufts Medical Center
Other Study IDs: 4530
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2006-10

CONDITIONS: Chronic Kidney Disease
Keywords: kidney disease; uric acid; outcomes; cardiovascular; mortality; kidney failure; Uric Acid levels in patients with Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non-diabetic Chronic Kidney disease

SUMMARY:
Patients in the earlier stages of Chronic kidney disease (CKD) are at risk both for the development of end-stage renal disease (ESRD) (define by the requirement for dialysis or kidney transplantation) and development of cardiovascular disease (CVD). Although controversial, there is literature to suggest that uric acid may play a role in the progression of kidney disease and development of cardiovascular disease (CVD). The Modification of Diet in Renal Disease (MDRD) Study was a randomized controlled trial in patients with CKD, which examined the effects of dietary protein restriction and strict blood pressure control on progression of non-diabetic CKD. Extensive data on risk factors for progression of kidney disease and development of CVD are available, as is long term follow up. 838 of the 840 patients who were randomized have uric acid levels measured at baseline. The aims of the present study are to examine the determinants of uric acid in cross sectional analysis at baseline, to determine the association between uric acid and development of ESRD, and the association of uric acid with all-cause and CVD mortality.

Level of kidney function will be a major determinant of uric acid levels independent of other risk factors.

Level of uric acid will be associated with development of ESRD independent of level of kidney function and other risk factors.

Uric Acid levels will be associated with both all-cause and CVD mortality independent of kidney function and other risk factors.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years of age
* with serum creatinine of 1.2 to 7 mg/dl in women and 1.4 to 7 mg/dl in men

Exclusion Criteria:

* pregnancy
* Type I diabetes
* insulin dependent type II diabetes
* renal artery stenosis
* proteinuria greater than 10mg/day
* mean arterial pressure greater than 125 mmHg
* prior kidney transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 838 participants of the randomized arm of the Modification of Diet in Renal Disaese (MDRD) Study conducted between 1989-1993
Sampling Method: Non-Probability Sample
Enrollment: 838 (Actual)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Kidney Failure

SECONDARY OUTCOMES:
CVD and All-Cause Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States